CLINICAL TRIAL: NCT04445116
Title: A Study of Endeavor™, a Video-Game Based Cognitive Remediation, in the Pediatric Multiple Sclerosis (MS) Population
Brief Title: Endeavor™ in Pediatric MS
Acronym: Akili
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funds and limited staffing to complete the pilot program.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-00634
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Endeavor™ Action Video Game Treatment (Experimental): 25 participants will fill out questionnaires and complete a neuropsychological evaluation. During study participation, participants will target using Endeavor™ action video game to complete 25-30 minutes at-home sessions 5 days a week for a total of 8 weeks via an iOS application.
  Interventions: Device: Action Video Game Treatment

INTERVENTIONS:
Device: Action Video Game Treatment — Endeavor™ is a digital, non-drug investigational treatment that is delivered through an action video game and is designed to target cognitive deficits in adolescence and young adults with pediatric onset MS.
  Other Names: Endeavor™

SUMMARY:
This study will examine the feasibility of using an Endeavor™ application as a treatment modality for cognitive impairments in the pediatric MS population. Participants will be asked to undergo a hour-long baseline evaluation, followed by at-home Endeavor™ application sessions. Subjects will complete the User Experience Feedback Form weekly on REDCap and at the end of the study. They will undergo another hour-long follow-up evaluation at the end of the study.

DETAILED DESCRIPTION:
Duration of subject participation in this study is anticipated to take 3-4 months. After consent/assent, participants will complete an one hour-long baseline study visit in-person at the MSCCC, or through a video visit. During this visit, participants will complete a neuropsychological evaluation and baseline study surveys and get trained on the use of the Endeavor™ video game. Participants will then be instructed to target a completion of at-home game play 5 days a week, for a total period of 8 weeks, using their own iOS mobile device, or a study-provided device if needed, approximately 25-30 minutes each day. Subjects will be instructed to complete the User Experience Feedback Form weekly via REDCap to assess feasibility and acceptability of Endeavor™. At the conclusion of participation, participants will complete an hour long neuropsychological evaluation and end of study User Experience Feedback Form via REDCap (in-person at the MSCCC, or through a telehealth video visit).

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment: 12 years 0 months to 22 years 11 months
* Confirmed Diagnosis of Multiple Sclerosis with onset < 17 years and 11 months (defined by the 2013 International Pediatric MS Study Group (IPMSSG) criteria (Krupp, Tardieu, Amato, Banwell, Chitnis, Dale, Ghezzi, Hintzen, Kornberg, Pohl, Rostasy, Tenembaum, Wassmer, & Sclerosis, 2013) and the 2010 McDonald criteria (Polman et al., 2011).)
* Followed at NYU Langone Health MSCCC
* Expanded Disability Status Scale (EDSS) score of ≤3.5

Exclusion Criteria:

* Previous report of an IQ < 70
* Non-English speaking, learned English in the past three years, or learned English after the age of 12 years
* Neurological disorder (other than MS) with potential to significantly influence cognition (e.g. head injury)
* Other serious chronic or unstable medical condition (e.g., epilepsy, sickle cell disease, Type 1 diabetes)
* Not willing to comply with all study procedures
* Insufficient visual and motor ability to carry out academic and cognitive tests
* Relapse ≤ 2months prior to academic and cognitive data collection
* Steroid treatment ≤ 1 month prior to academic and cognitive data collection

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Percent compliance for total at-home sessions | End of study (Day 60)
  Participants will be categorized as "compliant" if they interact with the mobile Endeavor™ a minimum of 3 times per week for a minimum of six of the eight weeks across the study period of 60 days.

SECONDARY OUTCOMES:
Change in Fatigue in Adult participants | Baseline (Day 0), End of study (Day 60)
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue form will be completed by the adult MS patients (7 questions). The PROMIS Fatigue instrument evaluate a range of self-reported symptoms that likely decrease the subjects' ability to carry out daily activities and might have an influence on cognitive function and processing speed.
Change in Fatigue in Pediatric participants | Baseline (Day 0), End of study (Day 60)
  The PROMIS Pediatric Fatigue form (23 questions) will be completed by the pediatric MS subjects enrolled in this study. The PROMIS Fatigue instrument evaluate a range of self-reported symptoms that likely decrease the subjects' ability to carry out daily activities and might have an influence on cognitive function and processing speed.
Change in Depression in Participants | Baseline (Day 0), End of study (Day 60)
  The PROMIS Depression form (28 questions) and PROMIS Pediatric Depression form (13 questions) evaluates self-reported negative mood symptoms and social cognition. This assessment will be completed for the adult MS patients (PROMIS Depression) and the pediatric MS subjects (PROMIS Pediatric Depression).
Change in Quality of life in Participants | Baseline (Day 0), End of study (Day 60)
  The MS Quality of Life Inventory (MSQoL) 54 Instrument is a health-related quality of life measure that combines both generic and MS-specific items and will be completed by the adult MS patients enrolled in this study. The instrument consists of 54 self-report items and yields two summaries, a health composite summary and a mental health composite summary.
Change in behaviors in pediatric participants. | Baseline (Day 0), End of study (Day 60)
  To determine and control for depressive and other behavioral symptoms on cognitive functioning, the Behavioral Assessment Scale for Children Third Edition (BASC-III) will be administered to pediatric MS subjects in this study. The assessments describe specific behaviors that are rated on a four-point scale of frequency, ranging from Never to Almost Always and include statements such as "My parents listen to what I say" and "I like to take risks." This 189-item assessment will help in determining behavioral patterns. These rating scales are performed on a computer.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health - Ambulatory Care Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. equests should be directed to leigh.charvet@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.